CLINICAL TRIAL: NCT04110119
Title: Effectiveness of Chiropractic Application in Patients With Acute Low Back Pain Presenting to the Emergency Department and Receiving Drug Treatment
Brief Title: Effectiveness of Chiropractic Application for Acute Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, ALI TIMUCIN ATAYOGLU, Assistant Prof., Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMUEC441
Record Dates: First submitted 2019-09-21; First posted 2019-10-01 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Low Back Pain, Mechanical
Keywords: Mechanical Low Back Pain; Chiropractics; Analgesic-anti-inflammatory; myorelaxant; Thiocolchicoside
MeSH Terms: conditions — Low Back Pain | interventions — thiocolchicoside

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control: Drug-Only Group (Active Comparator): Patients with acute lower-back pain who have undergone routine conventional drug treatment at the first visit to the emergency department (49 patients). The drug treatment consists of analgesic-anti-inflammatory (diclophenac sodium 75 mg IM) and myorelaxant (thiocolchicoside 4 mg IM), administered only once.
  Interventions: Drug: diclophenac sodium (75 mg, IM) and thiocolchicoside (4 mg, IM)
- Case: Drug and Chiropractic Group (Experimental): Patients, who received chiropractic treatment immediately after the conventional drug treatment as in the control group (49 patients). The chiropractic treatment consists of high speed and low amplitude spinal manipulation techniques, applied only once.
  Interventions: Drug: diclophenac sodium (75 mg, IM) and thiocolchicoside (4 mg, IM); Other: Chiropractic Treatment

INTERVENTIONS:
Drug: diclophenac sodium (75 mg, IM) and thiocolchicoside (4 mg, IM) — Single intramuscular injection of mixture of two commercial drugs (Analgesic-anti-inflammatory and myorelaxant) at the specified dosages
Other: Chiropractic Treatment — High speed and low amplitude spinal manipulation techniques are applied to the case group.
  Arms: Case: Drug and Chiropractic Group

SUMMARY:
The aim of this project is to investigate the effectiveness of chiropractic application on patients who have undergone routine medication as a standard hospital treatment for mechanical low-back pain as described in the Clinical Practice Guidelines

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 65.
* Acute lower-back pain, persisting less than 6 weeks, meeting the diagnostic classification of 1 or 2 according to the Quebec Task Force on Spinal Disorders

Exclusion Criteria:

* Previous spine surgery
* Spinal nerve root irritation or deficits,
* Pregnant women,
* Lower-back pain due to occupational accidents
* Obesity status (body mass index> 30).
* Chronic lower-back pain longer than 6 weeks.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in pain level | Up to 5 minutes
  Visual Analogue Pain Scale (VAS) assessment at the fifth minute after the injection of drug. Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It uses a ten centimeter scale with a minimum of 0 indicating no pain and a maximum of 10 indicating worst pain.
Change in pain level | Up to 30 minutes
  Visual Analogue Pain Scale (VAS) assessment at the fifth minute after the injection of drug. Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It uses a ten centimeter scale with a minimum of 0 indicating no pain and a maximum of 10 indicating worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Beykoz, Istanbul, Turkey (Türkiye)